CLINICAL TRIAL: NCT03792126
Title: A Pilot Cluster Randomised Controlled Trial, of an Implicit Learning Approach (ILA) Versus Standard Care, on Recovery of Mobility Following Stroke
Brief Title: Implicit Learning in Stroke Study
Acronym: IMPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Bournemouth Hospital (Other)
Collaborators: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICA-CL-2017-03-011
Record Dates: First submitted 2018-12-19; First posted 2019-01-03 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Standard care, as per usual working practice for the stroke unit. Control stroke units will have minimal contact with the research team, other than for data collection. They will be aware of the broad aims of the study, but not the specific detail of the intervention.
- Implicit Learning Approach (Experimental): All mobility focussed rehabilitation sessions will utilise the Implicit Learning approach (ILA), as usual care. This includes rehabilitation (delivered by a physiotherapist, occupational therapist or therapy assistant) that focusses on sitting, sit to stand, standing, stepping, transfers and walking. The content of therapy will be based on the treatment guidelines and intervention manual, which have been developed by an international expert group (using Delhi methodology). As this is a clinically grounded, pragmatic trial, therapists will have freedom to tailor the specific content of each treatment session to patient need, whilst remaining true to the ILA. Other therapy interventions, such as upper limb rehabilitation, will be provided as usual.
  Interventions: Other: Implicit Learning Approach

INTERVENTIONS:
Other: Implicit Learning Approach — All mobility focussed rehabilitation sessions will utilise the Implicit Learning Approach (ILA), as usual care. This includes rehabilitation (delivered by a physiotherapist, occupational therapist or therapy assistant) that focusses on sitting, sit to stand, standing, stepping, transfers and walking. The content of therapy will be based on the treatment guidelines and intervention manual - and primarily involves changing the quantity and focus of attention of instructions and feedback.
  As this is a clinically grounded, pragmatic trial, therapists will have freedom to tailor the specific content of each treatment session to patient need, whilst remaining true to the ILA.
  Arms: Implicit Learning Approach

SUMMARY:
This trial will compare an Implicit Learning Approach (ILA) to usual care, during the rehabilitation of mobility post stroke.

It is a multicentre, assessor blind, cluster randomised controlled pilot trial, with embedded feasibility study. It also includes a nested qualitative evaluation, designed to explore the views of participants and therapists.

DETAILED DESCRIPTION:
Re-gaining the ability to stand, step and walk are common goals for people with stroke. During rehabilitation, therapists often tell people how to move, e.g. "straighten your knee when you're standing", or "lift your foot as you step". However, these types of specific instructions may not help people to learn new skills. Reducing the number of instructions or using simpler instructions may help people to learn in a more automatic way - e.g. through trial and error. This is called implicit learning.

There is very little evidence into implicit learning in stroke. This study will investigate whether patients recover the ability stand, step and walk following stroke better when they are given fewer and simpler instructions.

We will do this using a cluster randomised design. We will invite up to 8 stroke units to take part - half will continue to deliver usual rehabilitation, and half will adopt an Implicit Learning Approach (ILA) for the duration of the trial. Which one of the two approaches the unit delivers will be chosen at random. At the ILA sites, therapists will be trained to deliver rehabilitation using fewer and less complex instructions.

All patients at each unit will receive their rehabilitation using the allocated approach. This helps to ensure that the therapy teams manage to deliver the interventions effectively. We will ask individual patients for permission to complete additional assessments, which form part of the study. Some participants and clinicians will be interviewed at the end of the study, to find out what they thought about the intervention.

This is a pilot study, meaning that we are testing how well this works as a research method. We will not know for certain which approach is best, but it will tell us how we should design a larger trial that will give a clear answer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke, presenting with hemiplegia
* Within 14 days of stroke onset
* Medically stable
* Able to...

  * tolerate daily therapy for a minimum of 30 minutes per session
  * sit for more than 5 seconds without support
  * understand and follow 1 stage commands

Exclusion Criteria:

* Previous stroke with residual impairments
* Other neurological diagnosis (e.g. Parkinsons Disease, Multiple Sclerosis)
* Clinically relevant pre-morbid disability levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise Johnson, Principal Investigator — University Hospitals Dorset
Locations (1):
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualitative data has been shared via the publication with PlosOne, as part of their publishing requirements. Quantitative data will be made available, upon reasonable request, following publication of the final paper.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Following final paper publication and for the duration of the archiving period (10 years)
Access Criteria: Will be assessed upon request.

REFERENCES:
- [Derived] Johnson L, Mardo J, Demain S. Understanding implementation of a complex intervention in a stroke rehabilitation research trial: A qualitative evaluation using Normalisation Process Theory. PLoS One. 2023 Sep 8;18(9):e0282612. doi: 10.1371/journal.pone.0282612. eCollection 2023. PMID 37682841
- [Derived] Johnson L, Burridge J, Ewings S, Westcott E, Gayton M, Demain S. Principles into Practice: An Observational Study of Physiotherapists use of Motor Learning Principles in Stroke Rehabilitation. Physiotherapy. 2023 Mar;118:20-30. doi: 10.1016/j.physio.2022.06.002. Epub 2022 Jun 20. PMID 36306569
- [Derived] Johnson L, Burridge J, Demain S, Ewings S. Comparing the Impact of an Implicit Learning Approach With Standard Care on Recovery of Mobility Following Stroke: Protocol for a Pilot Cluster Randomized Controlled Trial. JMIR Res Protoc. 2019 Nov 5;8(11):e14222. doi: 10.2196/14222. PMID 31687935

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Care: Standard care clusters will not have access to the trial materials (e.g. treatment manual), or details about the specific elements of the intervention.
Period: Overall Study
Arm/Group | Standard Care | Implicit Learning Approach
Started | 30 | 24
Completed | 27 | 14
Not Completed | 3 | 10
Not completed — Adverse Event | 1 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — COVID-19 Restrictions | 1 | 3
Not completed — Symptoms resolved | 0 | 3

BASELINE CHARACTERISTICS:
Population: 3 participants had withdrawn from the Implicit Learning Cohort prior to intervention starting due to symptom resolution and were not therefore included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Implicit Learning Approach | Total
Number analyzed (Participants) | 30 | 21 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (15) | 73 (12) | 74 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 7 | 22
  Male | 15 | 14 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 30 | 21 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Rivermead Mobility Index Score
Description: Measure of functional mobility in people with stroke.
  Ordinal scale, measured through direct observation of function.
  Score range from 0-40, with a higher score indicating better functional mobility status.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Implicit Learning Approach
Number analyzed (Participants) | 27 | 14
score on a scale | 30.2 (11.6) | 34.4 (7.5)

2. Secondary Outcome: Swedish Postural Adjustment in Stroke Scale (SwePASS)
Description: Measure of postural control in people with stroke, from lying, sitting and standing postures.
  Ordinal scale, measured through direct observation of function.
  Score range from 0-36, with a higher score indicating better postural control.
Time Frame: Week 0, 2 and 12
Population: Patients had withdrawn over at each time point in both interventions for different reasons including 2 further stroke, 1 did not attend, 5 affected by COVID-19 restrictions, 1 death and 1 patient choice withdrawal. 3 participants withdrew prior to the start of the intervention in the implicit learning approach as their symptoms had resolved, therefore they were not included in analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Care | Implicit Learning Approach
Number analyzed (Participants) | 30 | 21
units on a scale
  Week 0 | 17.7 (6.2) | 19.3 (7.5)
  Week 2: number analyzed (Participants) | 29 | 18
  Week 2 | 22.1 (6.8) | 23.9 (8.1)
  Week 12: number analyzed (Participants) | 27 | 14
  Week 12 | 26.4 (7.8) | 29.1 (5.3)

3. Other Pre Specified Outcome: Fugl Meyer - Motor Leg Sub Section
Description: Measure of sensori-motor function in the lower limb (impairment level)
  Range 0-28, with higher score indicating better outcome.
Time Frame: Week 0, week 2 and week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Implicit Learning Approach
Number analyzed (Participants) | 30 | 21
score on a scale
  Week 0 | 14.0 (7.6) | 11.5 (7.0)
  Week 2: number analyzed (Participants) | 29 | 18
  Week 2 | 17.65 (7.2) | 16.3 (9.7)
  Week 12: number analyzed (Participants) | 27 | 14
  Week 12 | 21.1 (8.0) | 24.9 (6.0)

4. Other Pre Specified Outcome: Modified Rankin Score
Description: Measure of disability and dependence in people who have suffered a stroke.
  Score 0-6, with higher score indicating a worse outcome.
Time Frame: Week 0, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Implicit Learning Approach
Number analyzed (Participants) | 30 | 21
score on a scale
  Week 0 | 4 (0) | 3.96 (0.21)
  Week 12: number analyzed (Participants) | 27 | 14
  Week 12 | 4 (0.9) | 2.6 (1.0)

5. Other Pre Specified Outcome: EuroQOL 5 D Questionnaire Index Score
Description: Standardised self-administered questionnaire to measure health related quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored based on the participant ticking the statement that best fits them. The statements range from "I have no problems..." to "I am unable to..." and are given a score 1-5 with a total score being between 5 and 25. Higher score indicates a worse outcome.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Implicit Learning Approach
Number analyzed (Participants) | 27 | 14
score on a scale | 12 (4) | 13.2 (4)

ADVERSE EVENTS:
Time Frame: Serious Adverse events data were collected from consent until end of trial intervention period (discharge from hospital - an average of 31 days for control group and 34 days for intervention group).
Description: 3 participants withdrew prior to the start of the intervention in the implicit learning approach as their symptoms had resolved, therefore they were not included in analysis.
Arm/Group | Standard Care | Implicit Learning Approach
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/21
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/21
Other Adverse Events (participants affected / at risk) | 0/30 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Care (N=30) | Implicit Learning Approach (N=21)
Stroke (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03792126/Prot_SAP_000.pdf